CLINICAL TRIAL: NCT05400031
Title: Does Oral Care With Propolis Affect the Development of Oral Mucositis in Pediatric Oncology Patients: A Randomized Controlled Clinical Study
Brief Title: Oral Care With Propolis in Pediatric Oncology Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Collaborators: Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Beste Ozguven Oztornaci, Asst. Prof., Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022/61
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Oral Mucositis
MeSH Terms: conditions — Stomatitis | interventions — Propolis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): In this group, the researcher will provide the participants with routine care.
- placebo group (Placebo Comparator): In this group, the researcher will provide the participants with a propolis vehicle
  Interventions: Biological: Placebo
- propolis group (Active Comparator): In this group, the researcher will provide the participants with a propolis solution.
  Interventions: Biological: propolis

INTERVENTIONS:
Biological: propolis — After obtaining written consent, oral identification of all participants will be performed prior to randomization. Oral diagnosis of children receiving chemotherapy will be repeated on day 0, day 5, and day 10, and the difference between the Oral Mucositis Rating Scale mean scores of the children in the groups will be examined.
  Oral Mucositis Assessment: Oral Mucositis Rating Scale will be used. The oral mucosa of children will be evaluated using the World Health Organization Oral Mucositis Classification.
  Arms: propolis group
Biological: Placebo — Placebo
  Arms: placebo group

SUMMARY:
According to the data from the World Health Organization, approximately 14 million people are diagnosed with cancer every year, and this number is expected to increase further in the next 10 years. Multidisciplinary treatment consisting of chemotherapy, radiotherapy and surgery is applied in childhood cancers. In chemotherapy, the target is cancerous cells, but high doses of chemotherapeutic agents do not have selectivity. Intact tissue cells are also affected by this cytotoxicity. Mucositis develops in the patient, especially as a result of the mucosal cells being affected. Mucositis is defined as damage to the mucosa lining the oral cavity, pharynx, larynx, oesophagus and gastrointestinal tract due to cancer treatment. It is one of the most important side effects of both chemotherapy and radiotherapy. This study is carried out to determine the effectiveness of propolis in preventing the formation of oral mucositis due to multiple use of chemotherapeutic drugs.

DETAILED DESCRIPTION:
According to the data from the World Health Organization, approximately 14 million people are diagnosed with cancer every year, and this number is expected to increase further in the next 10 years. Multidisciplinary treatment consisting of chemotherapy, radiotherapy and surgery is applied in childhood cancers. In chemotherapy, the target is cancerous cells, but high doses of chemotherapeutic agents do not have selectivity. Intact tissue cells are also affected by this cytotoxicity. Mucositis develops in the patient, especially as a result of the mucosal cells being affected. Mucositis is defined as damage to the mucosa lining the oral cavity, pharynx, larynx, oesophagus and gastrointestinal tract due to cancer treatment. It is one of the most important side effects of both chemotherapy and radiotherapy. This study is carried out to determine the effectiveness of propolis in preventing the formation of oral mucositis due to multiple uses of chemotherapeutic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Receiving chemotherapy treatment for lymphoproliferative malignant disease (leukaemia, lymphoma) or other childhood solid tumour (such as central nervous system tumour, neuroblastoma, osteosarcoma, Ewing sarcoma, rhabdomyosarcoma, hepatoblastoma, germ cell tumours)
* Being between the ages of 2-18 (Although there is no harm in using propolis, it is inconvenient for children under the age of 2 to use honey and its by-products due to botulism)
* No development of oral mucositis
* The child who does not smoke

Exclusion Criteria:

* The patient does not receive head and neck RT (increases the incidence of oral mucositis by 40%).
* The patient is allergic to bee products.
* Exclusion Criteria and Practices in this Case:
* Development of an allergic reaction to propolis (Applied oral care protocol is stopped, removed from the sample)
* Starting RT
* The child's need for MV support

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 108 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Oral mucositis grading | first day of the intervention
  Oral Mucositis Assessment Scale is a classification method accepted by the World Health Organization and used all over the world. It has standard clauses that will be interpreted in the same way by all people. However, in order to ignore the differences in interpretation, multi-research evaluation will be used in the first 20 observations and the consistency between the observers will be analyzed with Kappa analysis and the follow-ups will continue.
Oral mucositis grading | fifth day of the intervention
  Oral Mucositis Assessment Scale is a classification method accepted by the World Health Organization and used all over the world. It has standard clauses that will be interpreted in the same way by all people. However, in order to ignore the differences in interpretation, multi-research evaluation will be used in the first 20 observations and the consistency between the observers will be analyzed with Kappa analysis and the follow-ups will continue.
Oral mucositis grading | tenth day of the intervention
  Oral Mucositis Assessment Scale is a classification method accepted by the World Health Organization and used all over the world. It has standard clauses that will be interpreted in the same way by all people. However, in order to ignore the differences in interpretation, multi-research evaluation will be used in the first 20 observations and the consistency between the observers will be analyzed with Kappa analysis and the follow-ups will continue.

CONTACTS AND LOCATIONS:
Overall Officials: ZUHAL ONER SIVIS, MD, Study Chair — Tepecik Research and Training Hospital
Locations (1):
- Tepecik Research and Training Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be decided on demand.